CLINICAL TRIAL: NCT05055427
Title: Efficacy of Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang With Ginseng) on Mild and Moderate COVID-19 Patients: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Efficacy Evaluation of Shen Cao Gan Jiang Tang on Mild and Moderate COVID-19 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, NGUYEN VAN DAN, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 458/HĐĐĐ-ĐHYD
Record Dates: First submitted 2021-09-21; First posted 2021-09-24 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Respiratory Infection; Herbal Medicine
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, randomized controlled trial, we recruited patients with Covid-19 from five temporary for COVID-19 treatment in Ho Chi Minh City, Viet Nam.
  The protocol was designed based on the Good Clinical Practice guidelines and The Declaration of Helsinki. Number of Participants have 150 mild COVID-19 patient and 150 moderate COVID-19 patient. In each group of mild or moderate patients, we plan to randomize in a 1:1 ratio. Subjects in the investigational group will receive Shen Cao Gan Jiang Tang in addition to the Standard of Care (SOC) for the treatment of COVID-19 based on the Vietnam Ministry of Health guideline. Subjects in the controlled group will receive the Standard of Care (SOC) for the treatment of COVID-19 based on the Vietnam Ministry of Health guideline.
Masking Description: An open-label study was conducted because of the urgency of major public health events
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Experimental: Investigational arm (Experimental): Patients take Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) and the Standard of Care (SOC) for the treatment of COVID-19 based on the Vietnam Ministry of Health guideline.
  Interventions: Drug: Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng)
- • Controlled arm (No Intervention): Patients receive the Standard of Care (SOC) for the treatment of COVID-19 based on the Vietnam Ministry of Health guideline

INTERVENTIONS:
Drug: Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) — Patients take Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng), one bag of decoction (90ml) two times a day for 10 days. In additional, patients also receive the Standard of Care (SOC) for the treatment of COVID-19 based on the Vietnam Ministry of Health guideline.
  Ingredients per formula (tang): 12 grams of honey-fried Radix Glycyrrhizae, 6 grams of Rhizoma Zingiberis (stir-baked), 6 grams of Panax Ginseng. The decoction of concentrated extract is packed into aluminum foil vacuum bag, 90ml per bag, 1 formula (tang) is equivalent to 2 bags. Patients use the decoction directly from the bag.
  Daily dose: 1 bag per time, 2 times per day
  Other Names: "Sâm Thảo Can khương thang (Cam thảo Can khương gia Nhân sâm)"
  Arms: • Experimental: Investigational arm

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the virus that causes COVID-19 (coronavirus disease 2019). Patients with COVID-19 may experience various clinical manifestations, from no symptoms to critical illness such as severe pneumonia and acute respiratory distress syndrome (ADRS). So far, there is no specific medication for COVID-19; hence, the current available treatments mostly aim at symptoms management and supportive care. From traditional medicine perspective, COVID-19 is classified as warm-disease (Wen-yi). The main points of treatment for COVID-19 in early stage based on traditional medicine perspective are strengthen the Protective Qi (Wei Qi - the body immune system), and restore the balance of Qi, which is vital biological energy to prevent the invasion of external pathogens, including the SARS-CoV-2 virus. The Shen Cao Gan Jiang Tang have including Gan Cao Gan Jiang Tang (GGT) with the addition of Ginseng. This formula is originated from Shang Han Lun (Treatise on Febrile Diseases Caused by Cold) by Zhang Zhong-jing, used to enhance the Protective Qi, treat the early stage of Febrile Diseases, This clinical trial aims to evaluate the efficacy of the Shen Cao Gan Jiang Tang on mild and moderate COVID-19 patients

DETAILED DESCRIPTION:
The main objectives of this clinical trial:

1. Assess the efficacy of Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) in addition to the standard of care on reducing duration and severity of symptoms compared with the standard of care in mild and moderate COVID-19 patients.
2. Assess the efficacy of Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) in addition to the standard of care on reducing the proportion of patients progressed to severe level compared with the standard of care in mild and moderate COVID-19 patients.
3. Assess the efficacy of Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) in addition to the standard of care on reducing the time required to meet discharge standards compared with the standard of care in mild and moderate COVID-19 patients.

This study is investigated by the following hypotheses: combining Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) with the standard of care is effective in reducing the duration and severity of symptoms, reducing the proportion of patients progressed to severe level, and reducing the length of hospital stay on mild and moderate COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* From full 18 to 64 years old;
* The patient was diagnosed with SARS-CoV-2 infection by RT-PCR confirmation (+) and CT < 30.
* Patients classified as mild (acute upper respiratory tract infection): patients infected with SARS-CoV-2 early in the first 5 days from the time of having one of the non-specific clinical symptoms such as fever, cough dry, sore throat, stuffy nose, fatigue, headache, muscle pain, decreased taste, decreased sense of smell. And there are no signs of pneumonia or hypoxia, respiratory rate ≤ 20 times/min, Saturation of Peripheral Oxygen (SpO2) ≥ 96% when breathing air.
* Patients classified as moderate (Pneumonia): patients infected with SARS-CoV-2 in the first 10 days from the time of having one of the non-specific clinical symptoms, showing signs of pneumonia (fever, cough, dyspnea, tachypnea >20 breaths/min) and no signs of severe pneumonia, Saturation of Peripheral Oxygen (SpO2) ≥ 93% when breathing air.
* Inpatient treatment
* Subjects do not use any other medicines with herbal ingredients for underlying conditions or any other purposes;
* Voluntary participation in the study by signing an informed consent
* Patients who have not been vaccinated or have just received 1 dose of COVID-19 vaccine

Exclusion Criteria:

* Severe or critical COVID-19 based on the COVID-19 severity scale of Vietnam Ministry of Health;
* Chronic obstructive pulmonary disease, kidney failure requiring dialysis or creatinine ≥ 2.0mg/dl through medical history; parenteral or parenteral nutrition, uncontrolled type 2 diabetes (HbA1c > 7%), uncontrolled hypertension (value > 160/100 mmHg), uncontrolled coronary artery disease (new/currently established) requires medication adjustment), heart failure, neurological disease (eg, acute stroke, polyneuritis within 1 month) or mental illness, active tuberculosis, active autoimmune disease;
* Have a chronically weakened immune system (AIDS, cancer, undergoing chemotherapy-radiotherapy in the past six months, immunosuppressive disease);
* Taking immunosuppressive drugs (e.g., anti-rejection treatment after organ transplant or blood stem cell transplant);
* Allergic to products that contain ginseng;
* Pregnant or lactating women;
* Already participating in another clinical trial;
* The patient has received 2 doses of COVID-19 vaccine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Duration of symptoms of COVID-19 | From Day 1 to Day 21 after randomization
  Time (days) from randomization to symptoms disappear
The severity of the COVID-19 total and individual symptoms | From Day 1 to Day 21 after randomization
  Time (days) from randomization to the relief of total and individual COVID-19 symptoms scores
Rate of progression to disease severity | During inpatient treatment, maximum to Day 21 after randomization
  Number of patients (%) progressed to severe level of COVID-19 severity scale based on the Vietnam Ministry of Health severity scale during the period of the treatment
The time required to meet discharge standards | During inpatient treatment, maximum to Day 21 after randomization
  Time (days) from randomization to get required for a negative real-time polymerase chain reaction (RT-PCR) testing for SARS-CoV-2 or CT > 30
National Early Warning Score 2 (NEWS2) | During inpatient treatment, maximum to Day 21 after randomization
  Assessed by National Early Warning Score 2 (NEWS2)

SECONDARY OUTCOMES:
Cycle threshold (CT) | During inpatient treatment, maximum to Day 21 after randomization
  Cycle threshold (CT) values on the COVID-19 RT-PCR test
Duration of SARS-CoV-2 virus infection | During inpatient treatment, maximum to Day 21 after randomization
  Time (days) from randomization to negative the COVID-19 RT-PCR test
Mortality rate | From Day 1 to Day 21 after randomization
  The number of deaths (%) caused by COVID-19
Number of participants clinically recovered | From Day 1 after randomisation to Day for patients meet discharge criteria
  Number of patients (n) without symptoms of COVID-19 on date of discharge
Paracetamol/Ibuprofen intake | From Day 1 after randomisation to Day for patients meet discharge criteria
  The number (n) of daily doses of paracetamol/ibuprofen consumed during inpatient
Safety evaluation | From Day 1 to Day 21 after randomization
  Number of patients (n) that have the side effects due to the decoction based on clinical monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Van-Dan Nguyen, MD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No